CLINICAL TRIAL: NCT02746536
Title: Effects of Slow Chest Compression on Dynamic Hyperinflation, Dyspnea and Peripheral Muscle Deoxygenation Induced by Exercise in Patients With COPD
Brief Title: Slow Chest Compression on Dynamic Hyperinflation, Dyspnea and Peripheral Muscle Deoxygenation in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Prof. Dra. Anamaria Fleig Mayer, PhD, University of the State of Santa Catarina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SCC2016
Record Dates: First submitted 2016-04-08; First posted 2016-04-21 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Inspiratory capacity; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slow chest compression (Experimental): Patients will receive the slow chest compression for one minute, immediately after 6MST.
  Interventions: Other: Slow chest compression
- No slow chest compression (Placebo Comparator): Immediately after 6MST, the patient will not receive the SCC and will remain seated at rest for one minute, without any intervention.
  Interventions: Other: No slow chest compression

INTERVENTIONS:
Other: Slow chest compression — During the SCC, the patient will remain in the sitting position; a bimanual slow compression on his/her upper chest will be performed always by the same evaluator, who will stand behind the patient. This compression will be done only in the expiratory phase, during one minute, in all respiratory cycles, respecting the chest mobility of each patient.
  A standardized verbal command will be given: "Exhale all the air".
  Arms: Slow chest compression
Other: No slow chest compression — The patient will remain seated at rest for one minute after the 6MST. A standardized verbal command will be given: "Exhale all the air".
  Arms: No slow chest compression

SUMMARY:
Background: Commonly, patients with chronic obstructive pulmonary disease (COPD) present dyspnea, dynamic hyperinflation (DH) and important peripheral muscle deoxygenation when performing their activities of daily living (ADLs). The slow chest compression (SCC) technique is a physiotherapy strategy that could maybe reduce DH, dyspnea and peripheral muscle deoxygenation in patients with COPD. The aim of the study is to analyse the effects of SCC in DH, dyspnea and peripheral muscle deoxygenation induced by exercise tests. The secondary objective was to identify responders and non-responders to the technique.

Design: Randomized cross-over study. Setting: The study will be conducted in an outpatient pulmonary rehabilitation program in Florianopolis, Brazil

Subjects: Patients with COPD (GOLD 2-4).

Interventions: Patients will randomly receive or not the SCC after six-minute step test (6MST-SCC and 6MST-NonSCC).

Main measures: At baseline and 1 minute after the tests, the inspiratory capacity (IC) will be assessed by the slow vital capacity (SVC) maneuver. At baseline, immediately after, and 1 minute after the tests, the dyspnea score will be assessed. The physiological responses and the peripheral muscle deoxygenation will be assessed during the tests and 1 minute after them.

DETAILED DESCRIPTION:
The period from August 2015 to April 2016 was designated to clinical trial design and to its submission/approval by the Human Research Ethics Committee. The recruitment of subjects and the study evaluations following described will be only initiated after registration and publication on the ClinicalTrials.gov platform.

Pulmonary function tests:

* Lung function will be tested using a total body plethysmography (Eric Jaeger, Germany), and the calibration will be checked before each evaluation. Spirometry will be performed in accordance with American Thoracic Society and European Respiratory Society (ATS/ERS) standards (Miller et al., 2005; Wanger et al., 2005). The predicted values will be calculated with the equations derived from Brazilian population (Pereira et al., 2007; Neder et al., 1999).
* SVC maneuver: IC will be measured with the patient in the sitting position, using a portable spirometer (NDD Medical Technologies®, Switzerland), before and 1 minute after the tests, by the SVC maneuver starting from a stable end-expiratory volume, in accordance with ATS/ERS standards (Miller et al.,2005). A minimum of three maneuvers (maximum of eight) will be performed and, in order to be considered reliable, two curves could not vary more than 5% or 150 ml. The higher value of two reproducible curves will be used for analysis (O'Donnell et al., 2001). This outcome will be collected by a third evaluator blinded for the SCC or non-SCC application.

Six-minute step test (6MST): The patients will be instructed to walk up and down the step in order to perform the largest number of steps during six minutes. The walking speed will be selected by the patient (da Costa et al., 2014;. Pessoa et al., 2014). Two 6MSTs will be conducted by two evaluators: the main evaluator will be responsible for conducting the tests and the other will count the number of steps performed by the patient.

Dyspnea: Before and after the completion of each 6MST and each 6MWT, patients will be asked about their perception of dyspnea, using the modified Borg scale. Immediately after completion the SCC (or not), patients will be asked again about the dyspnea score. This outcome will be collected by a third evaluator blinded for the SCC or non-SCC application.

Peripheral muscle oxygenation: During the tests, before and after the completion of each 6MST, it will be measured the peripheral muscle oxygenation by near-infrared spectroscopy (NIRS) (Artinis Medical Systems®, Netherlands). The device will be positioned over the vastus lateralis muscle of dominant leg.

Slow chest compression: The patient will receive in a randomized order the application or not of SCC for one minute immediately after 6MST. During the SCC, the patient will remain in the sitting position; a bimanual slow compression on his/her upper chest will be performed always by the same evaluator, who will stand behind the patient. This compression will be done only in the expiratory phase, during one minute, in all respiratory cycles, respecting the chest mobility of each patient. For all patients, during SCC, it will be given a standardized verbal command: "Exhale all the air". After the test in which the patient will not receive the SCC, he/she must remain seated, at rest, for one minute without any interventions, although it will be given the same standardized verbal command.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD confirmed by spirometry (COPD GOLD stages B, C and D)
* Absence of change in respiratory symptoms in the past four weeks
* No hospital admission in the past 12 weeks
* Age between 40 and 80 years-old

Exclusion Criteria:

* Any other disease or health condition that could compromise the test´s execution
* Participation in pulmonary rehabilitation program completed in the last six months
* Current smoking or its cessation in less than six months
* Any change in symptoms during the study protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Patients with COPD will perform the inspiratory capacity (IC) by the slow vital capacity (SVC) maneuver in order to measure dynamic hyperinflation (DH). | Change from baseline and exactly 1 minute after the 6MST and 6MWT
  Dynamic hyperinflation will be considered an increase of 150 ml or 10% on EELV after 6MST and 6MWT. End-expiratory lung volume (EELV) will be measured by the difference between total lung capacity and IC.
Patients with COPD will answer dyspnea score by modified Borg scale | Change from baseline, after the completion of each 6MST and 6MWT and exactly 1 minute after the SCC or non-SCC.
Patients with COPD will be monitored regarding peripheral muscle oxygenation by the near-infrared spectroscopy | Change from baseline, after the completion of each 6MST and 6MWT and exactly 1 minute after the SCC or non-SCC.

CONTACTS AND LOCATIONS:
Overall Officials: Anamaria F Mayer, PhD, Study Director — University of the State of Santa Catarina
Locations (1):
- Núcleo de Assistência, Ensino e Pesquisa em Reabilitação Pulmonar, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The autors declared that will be shared: individual deidentified participant data; individual data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices); Study Protocol, Statistical Analysis Plan, Informed Consent Form; immediately following publication and ending 5 years following article publication; With Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose to achieve aims in the approved proposal; proposals should be directed to anamaria.mayer@udesc.br to gain access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: immediately following publication and ending 5 years following article publication
Access Criteria: With Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose to achieve aims in the approved proposal; proposals should be directed to anamaria.mayer@udesc.br to gain access.

REFERENCES:
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Pereira CA, Sato T, Rodrigues SC. New reference values for forced spirometry in white adults in Brazil. J Bras Pneumol. 2007 Jul-Aug;33(4):397-406. doi: 10.1590/s1806-37132007000400008. English, Portuguese. PMID 17982531
- [Background] O'Donnell DE, Revill SM, Webb KA. Dynamic hyperinflation and exercise intolerance in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Sep 1;164(5):770-7. doi: 10.1164/ajrccm.164.5.2012122. PMID 11549531
- [Background] Wanger J, Clausen JL, Coates A, Pedersen OF, Brusasco V, Burgos F, Casaburi R, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson D, Macintyre N, McKay R, Miller MR, Navajas D, Pellegrino R, Viegi G. Standardisation of the measurement of lung volumes. Eur Respir J. 2005 Sep;26(3):511-22. doi: 10.1183/09031936.05.00035005. No abstract available. PMID 16135736
- [Background] Neder JA, Andreoni S, Castelo-Filho A, Nery LE. Reference values for lung function tests. I. Static volumes. Braz J Med Biol Res. 1999 Jun;32(6):703-17. doi: 10.1590/s0100-879x1999000600006. PMID 10412549
- [Background] da Costa JN, Arcuri JF, Goncalves IL, Davi SF, Pessoa BV, Jamami M, Di Lorenzo VA. Reproducibility of cadence-free 6-minute step test in subjects with COPD. Respir Care. 2014 Apr;59(4):538-42. doi: 10.4187/respcare.02743. Epub 2013 Sep 17. PMID 24046461
- [Background] Pessoa BV, Arcuri JF, Labadessa IG, Costa JN, Sentanin AC, Di Lorenzo VA. Validity of the six-minute step test of free cadence in patients with chronic obstructive pulmonary disease. Braz J Phys Ther. 2014 May-Jun;18(3):228-36. doi: 10.1590/bjpt-rbf.2014.0041. PMID 25003275
- [Background] Singh SJ, Puhan MA, Andrianopoulos V, Hernandes NA, Mitchell KE, Hill CJ, Lee AL, Camillo CA, Troosters T, Spruit MA, Carlin BW, Wanger J, Pepin V, Saey D, Pitta F, Kaminsky DA, McCormack MC, MacIntyre N, Culver BH, Sciurba FC, Revill SM, Delafosse V, Holland AE. An official systematic review of the European Respiratory Society/American Thoracic Society: measurement properties of field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1447-78. doi: 10.1183/09031936.00150414. Epub 2014 Oct 30. PMID 25359356